CLINICAL TRIAL: NCT07204626
Title: Medical Anthropology and Migrants in Precarious Situations, Cared for in Intensive and Post-intensive Care Units
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0110_REANIMATION
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-05

CONDITIONS: Anthropology; Immigrant; Intensive Care (ICU); Precariousness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months

GROUPS / COHORTS (2):
- patient
- medical staff

SUMMARY:
Analyze the experience (perception, interpretation and incorporation - embodiment) that migrant people with low socio-economic status/precarity have of their own health conditions for which they have come to be hospitalized in the Intensive Care Unit (ICU) and Post-Resuscitation Rehabilitation Care (PRRC).

ELIGIBILITY:
Inclusion Criteria:

For patients:

Male and female migrants (born outside of France and its territories, regardless of date of arrival, length of residence, or acquired nationality)

Aged 18 years or older

Living in or transiting through France

With or without residence permits or legal documentation

Hospitalized in ICUs and receiving care in post-ICU rehabilitation units (SRPR)

Providing consent to participate in the study

Having good proficiency in French, Spanish, or Italian, or, if not, benefiting from professional interpretation (ISM) or cultural mediation ensuring effective communication

Having a psychological and neurological state compatible with providing informed consent and taking part in an interview

For healthcare professionals and associative actors:

Being a healthcare, social work, or associative professional

Involved in the medical, psycho-social, and/or legal support and care of migrant patients admitted to ICUs and SRPR

Providing consent to participate in the study

Exclusion Criteria:

For patients:

Being born in France

Being a minor (<18 years old)

Being under guardianship or curatorship

Having a neurological state incompatible with providing informed consent and taking part in an interview

For healthcare professionals and associative actors:

Not being involved in the care of migrant patients admitted to ICUs and SRPR

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult migrant patients (≥18 years old) hospitalized in intensive care units (ICU) and receiving post-ICU rehabilitation care (SRPR) in selected French hospitals (Saint-Denis, Gonesse, Avicenne, Bichat). Eligible patients include those born outside France, regardless of their date of arrival, length of residence, or nationality, and who are able to communicate in French, Spanish, or Italian, either directly or via professional interpretation or cultural mediation. Participants must have a psychological and neurological state compatible with providing informed consent and participating in interviews.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Exploration of the lived experience and perceptions of health and critical care among socio-economically vulnerable migrant patients hospitalized in intensive care units (ICU) and post-ICU rehabilitation units (SRPR), assessed through semi-structured int | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Saint-Denis, Saint-Denis, France, France